CLINICAL TRIAL: NCT02071017
Title: Application of the Simultaneous PET (FDG)-MR Imaging for the Adult Patients Presented With Brain Tumor From Differential Diagnosis to Prediction of Prognosis
Brief Title: PET (FDG)-MR Imaging for the Adult Patients Presented With Brain Tumor
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Hong Choi, Seoul National University Hospital, Seoul National University Hospital
Other Study IDs: D-1212-014-447
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background and purpose: In adult, the half of the CNS neoplasms are metastatic, and high grade astrocytomas and oligodendrogliomas are most frequent malignant tumors among the last half. Recently, integrated MRI-PET (Biograph mMR, Siemens, Germany) was introduced, and can provide simultaneous whole body MRI-PET imaging as well as brain-specific advanced imaging (e.g. DWI, PWI, and DCE). The purpose of the present study is to evaluate whether the simultaneous MRI-PET acquisition can improve the diagnostic yield for the patients initially presented with brain tumors, and predict the prognosis in the patients diagnosed with primary high graded astrocytoma or oligodendroglioma.

DETAILED DESCRIPTION:
Materials and methods: Simultaneous MRI-PET (FDG) will be prospectively obtained in patients (n = 60) initially presented with brain tumors by using integrated MRI-PET (Biograph mMR, Siemens, Germany). We will exclude the patients suspected to have benign brain tumors such as meningioma and schwannoma on previous imaging studies. We will use the imaging protocols including whole body MRI-PET and advanced brain tumor imaging (DWI, PWI and DCE). In addition, we will analyze the imaging parameters to see whether the enrolled tumors are primary brain tumors or metastatic, and evaluate the tumor grading efficiency and prognosis prediction for the patients with high grade astrocytomas or oligodendrogliomas.

Expected results: We expect that whole body MRI-PET is useful for the differential diagnosis of primary and metastatic brain tumors, and the multiparametric information from DWI, PWI, DCE and PET can be used for the tumor grading and prognosis prediction of the primary brain malignancies.

ELIGIBILITY:
Inclusion Criteria:

* We will inculude the enrolled tumors are primary brain tumors or metastatic, and evaluate the tumor grading efficiency and prognosis prediction for the patients with high grade astrocytomas or oligodendrogliomas.

Exclusion Criteria:

* We will exclude the patients suspected to have benign brain tumors such as meningioma and schwannoma on previous imaging studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary brain tumors or metastatic, and evaluate the tumor grading efficiency and prognosis prediction for the patients with high grade astrocytomas or oligodendrogliomas.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
PET (FDG)-MR Imaging for the Adult Patients Presented With Brain Tumor | 2year

CONTACTS AND LOCATIONS:
Overall Officials: SeungHong Choi, MD, PhD, Principal Investigator — Seoul National University Hospital(Radiology)
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea